CLINICAL TRIAL: NCT01762618
Title: Experimental Study of the Impact of a Structured Psychological Intervention Based on Group Therapy for Caregivers of Alzheimer's Patients.
Brief Title: Experimental Study of the Impact of a Group Therapy Psychological Intervention for Caregivers of Alzheimer's Disease Patients
Acronym: EMOCUIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMOCUIDA/FPM-0211
Record Dates: First submitted 2012-12-18; First posted 2013-01-08 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Psychological Support to Caregivers of Azlheimer's Patients
Keywords: Group Cognitive Behavior Therapy, Alzheimer's disease, Caregivers¡
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy Group (Experimental): 14 therapy sessions, once a week for one and a half hours.
  Interventions: Behavioral: Cognitive Behavioral Therapy Group
- Control Group (No Intervention): Social support for caregiver (through the social worker) as usual. The social worker gives information when they considered that there is a social economic risk or upon request by the caregiver.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy Group — Therapy Groups
  Other Names: 14 therapy sessions, once a week for one and a half hours.
  Arms: Cognitive Behavioral Therapy Group

SUMMARY:
A randomized controlled trial designed to test the effectiveness of a psychological intervention based on group therapy for the caregivers of Alzheimer's disease patients. The intervention consists of 14 sessions of a cognitive-behavioral psychological group therapy. This study aims to demonstrate that Alzheimer's patients' caregivers can benefit from group counseling, with an improvement in mood state, quality of life, perceived burden and a decrease in anxiety and depression. Two evaluations will be done: before the therapy sessions (basal) and when intervention is finished (final).

DETAILED DESCRIPTION:
The aim of this study is to conduct group therapy with Alzheimer's caregivers at three centers in the province of Barcelona: Hospital El Carme Badalona, Sanitary Center of Les Corts and Sarrià.

The therapy sessions are conducted by an expert in group therapy (from the sponsor Pasqual Maragall Foundation) and the social worker of each of the centers. The study takes place for four months and consists of weekly therapy sessions of an hour and a half each (14 sessions in total), based on cognitive and behavioral theory. The participants and the control group are evaluated at the beginning and at the end of the study in terms of mood, quality of life, anxiety and depression.

This study aims to demonstrate that Alzheimer's patient's caregivers can benefit from group counseling, resulting in an improvement in their emotional state, perceived burden, quality of life and a more positive attitude coping with the new situation.

ELIGIBILITY:
Inclusion Criteria:

* To be the principal caregiver of a person with Alzheimer's disease
* The patient has a possible or probable diagnosis of Alzheimer's disease made for an Accredited Dementia Unit.
* The patient score in the Global Deterioration Scale must be: 4, 5 or 6A.
* The caregiver must dedicate at least 5 hours a day or spend a significant part of his time to care-related tasks
* The caregiver must sign the Informed Consent

Exclusion Criteria:

* To receive a financial compensation for the care of the patient
* The caregiver or the patient has a psychiatric illness according to the DSM-IV TR, such that the investigator considers it might hinder the dynamics of the group and affect the objectives of the study
* Be receiving some type of formal counseling (conducted by a therapist

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in POMS Scale ("Profile of Mood States") | Pre-treatment and 4 weeks post treatment
  Change from baseline compared to the control and active arms using the Profile of Mood State (POMS) validated in structure and content for the Spanish language. This scale is a popular instrument for mood evaluation. It comprises 44 items (with a Likert response from 0 to 4), representing six conceptual dimensions: tension, depression,anger, vigour, fatigue and friendliness.

SECONDARY OUTCOMES:
Change from baseline compared to the control and active arms using the Martin and cols. scale to assess the overload level of the family caregivers of patients with probable or possible Alzheimer's disease or other advanced stage dementia. | Pre-treatment and 4 weeks post treatment
  Martin and cols. scale is an adaptation of the Zarit questionnaire to assess the overload level of the caregiver. It is a self administered questionnaire, with 22 items with each item scored from 1 ('none') to 5 ('nearly always').

OTHER OUTCOMES:
Change from baseline compared to the control and active arms using the SF-36 v2 (Short Form-36 Health Survey), a questionnaire that measures the Quality of Life related to Health. | Pre-treatment and 4 weeks post treatment
  The SF-36 has 36 items that assesse eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems); bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. This version of the instrument asks for participants to reply to questions according to how they have felt over the previous four weeks. The items use Likert-type scales, some with 3, 5 or 6 points.
Change from baseline compared to the control and active arms using the Hospital Anxiety and Depression Scale (HADS) | Pre-treatment and 4 weeks post treatment
  The HADS is a fourteen item scale with a Likert response from 0 to 3 that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Poudevida, PhD, Principal Investigator — Barcelonabeta Brain Research Center, Pasqual Maragall Foundation
Locations (3):
- Spain (3):
  - Hospital del Carme, Badalona, Barcelona
  - Primary Assistant Center Les Corts, Barcelona, Catalonia
  - Primary Assistant Center Sarrià, Barcelona, Catalonia

REFERENCES:
- See also: Links to Pasqual Maragall Foundation Web page — http://www.fpmaragall.org